CLINICAL TRIAL: NCT04580342
Title: Comparative Study Between Oral Ivabradine Versus Oral Propranolol for Induced Hypotension in Functional Endoscopic Sinus Surgery
Brief Title: Ivabradine Versus Propranolol for Induced Hypotension in Endoscopic Sinus Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed talaat ahmed aly (Other)
Responsible Party: Sponsor-Investigator, Ahmed talaat ahmed aly, clinical professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ivabradine versus propranolol
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Ivabradine; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine group (Experimental)
  Interventions: Drug: oral Ivabradine
- propranolol group (Experimental)
  Interventions: Drug: oral Propranolol

INTERVENTIONS:
Drug: oral Ivabradine — Ivabradine group will receive ivabradine 5mg PO in the evening and 1 hour before anesthetic induction
  Arms: Ivabradine group
Drug: oral Propranolol — propranolol group will receive propranolol 10 mg PO in the evening and 1 hour before anesthetic induction.
  Arms: propranolol group

SUMMARY:
the study is designed to compare the effect of addition of oral Ivabradine, propranolol to general anesthesia aimed reduction in blood loss during functional endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years.
* Patients of both genders.
* ASA grade I - II .

Exclusion Criteria:

* Patient refusal.
* Any contraindication to medication included in the study .
* Patients with allergy to medication included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
change in blood loss | immediately after the surgery
  Estimated blood loss in millilitres per hour is calculated by subtracting the volume of total irrigation used during the case from the total amount of fluid in the suction canister at the end of surgery in addition, pre-weighing and post-weighing of sponges and oropharyngeal packs were also done and dividing by surgical time in hours.
  assessment of blood loss by Boezaart and van der Merwe Grading System for bleeding during Endoscopic Sinus Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed T Ahmed, A professor, Principal Investigator — Assiut University
Locations (1):
- Ahmed Talaat Ahmed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No